CLINICAL TRIAL: NCT06419829
Title: The Impact of Targeted Physical Activity on Body Composition, Posture and Physical Fitness of People of Different Ages
Brief Title: Physical Activity, Posture and Body Composition in Ontogeny
Status: Active, not recruiting | Type: Observational
Sponsor: Wroclaw University of Health and Sport Sciences (Other)
Responsible Party: Principal Investigator, Agnieszka Chwalczynska, PhD, Associate Professor, Wroclaw University of Health and Sport Sciences
Other Study IDs: AChwalWUHSS
Record Dates: First submitted 2024-05-08; First posted 2024-05-17 (Actual); Last update posted 2024-05-17 (Actual); Status verified 2024-05

CONDITIONS: Pediatric Obesity; Postural Balance; Physical Activity
Keywords: overweight and obesity; body posture; children's activity and physical fitness; activity and physical fitness of seniors; physioprophylaxis for falls
MeSH Terms: conditions — Pediatric Obesity; Motor Activity; Overweight; Obesity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (6):
- Pediatric group: Pediatric group - children aged 0-3 years old, participating in physiotherapeutic visits carried out as part of the assessment of the child's psychomotor development
  Interventions: Other: psychoprophylactic program aimed at improving physical fitness; Diagnostic Test: assessment of body posture using the Kasperczyk method
- Pediatric older group: Pediatric older group - Children aged 3-6 years recruited as part of pre-school education
  Interventions: Other: psychoprophylactic program aimed at normalizing body weight through medical training; Other: psychoprophylactic program aimed at improving body posture; Other: psychoprophylactic program aimed at improving physical fitness; Diagnostic Test: Body composition assessment; Diagnostic Test: assessment of body posture using the Kasperczyk method; Diagnostic Test: Assessment of physical fitness; Diagnostic Test: Balance assessment
- School group: School group - Children aged 7-15 recruited as part of compulsory schooling at primary school level
  Interventions: Other: psychoprophylactic program aimed at normalizing body weight through medical training; Other: psychoprophylactic program aimed at improving body posture; Other: psychoprophylactic program aimed at improving physical fitness; Diagnostic Test: Body composition assessment; Diagnostic Test: assessment of body posture using the Kasperczyk method; Diagnostic Test: Assessment of physical fitness; Diagnostic Test: Balance assessment
- Youth group: Respondents aged 15-25 recruited as part of secondary education, taking into account age (secondary school, university, graduate school) and gender division
  Interventions: Other: psychoprophylactic program aimed at normalizing body weight through medical training; Other: psychoprophylactic program aimed at improving body posture; Other: psychoprophylactic program aimed at improving physical fitness; Diagnostic Test: Body composition assessment; Diagnostic Test: assessment of body posture using the Kasperczyk method; Diagnostic Test: Assessment of physical fitness; Diagnostic Test: Balance assessment
- Adult group: Adult group - Respondents aged 25-55
  Interventions: Other: psychoprophylactic program aimed at normalizing body weight through medical training; Other: psychoprophylactic program aimed at improving physical fitness; Diagnostic Test: Body composition assessment; Diagnostic Test: Assessment of physical fitness; Diagnostic Test: Balance assessment
- Senior group: Senior group - Tests at the age of over 55, in the case of women, the condition for inclusion in this group is the postmenopausal period
  Interventions: Other: psychoprophylactic program aimed at normalizing body weight through medical training; Other: psychoprophylactic program aimed at improving body posture; Other: psychoprophylactic program aimed at improving physical fitness; Diagnostic Test: Body composition assessment; Diagnostic Test: assessment of body posture using the Kasperczyk method; Diagnostic Test: Assessment of physical fitness; Diagnostic Test: Balance assessment

INTERVENTIONS:
Other: psychoprophylactic program aimed at normalizing body weight through medical training — Based on the assessment of body weight and composition, a 12-week physiophylactic program will be carried out, adapted to the age and gender of the subjects. The program will be carried out twice a week for 30 to 60 minutes (depending on the group). The basis of the program will be the implementation of exercises that reduce fat mass, increase the flexibility and productivity of muscle mass. The classes will be conducted as part of medical training with a training load increasing to at least 85% of HR Max.
  The project will include theoretical classes for parents, children and seniors on eating habits, a proper age-appropriate diet, diet changes depending on the subject's health condition and physical activity, and the impact of diet on the process of puberty, adulthood and aging.
  Groups: Adult group; Pediatric older group; School group; Senior group; Youth group
Other: psychoprophylactic program aimed at improving body posture — Based on the body posture assessment, a 12-week physiotherapy program will be carried out, adapted to the age and gender of the subjects. The program will be carried out twice a week for 30 to 60 minutes (depending on the group). The basis of the program will be the implementation of exercises that strengthen the muscle corset, reducing asymmetrical positioning, habitual and during the implementation of professional tasks. The classes will be conducted using medical training and resistance exercises.
  The project will include theoretical classes for parents on sitting habits, the importance of physical activity in a child's development, the selection of footwear...
  Groups: Pediatric older group; School group; Senior group; Youth group
Other: psychoprophylactic program aimed at improving physical fitness — Based on the assessment of physical fitness, a 12-week physiotherapy program will be carried out, adapted to the age and gender of the participants. The program will be carried out twice a week for 30 to 60 minutes (depending on the group). The basis of the program will be the implementation of exercises aimed at improving physical fitness, with particular emphasis on impaired motor skills. The classes will be conducted using functional training, resistance and stretching exercises, strengthening all muscle groups. In the case of children, special attention will be paid to the strength of the upper limbs, in the case of seniors, balance and coordination exercises will be introduced to improve time and space orientation. In all groups, the main goal is to improve functional fitness The project will include theoretical classes for parents, children and seniors on the importance of physical activity in the quality of life, in the process of maturation and aging.
Diagnostic Test: Body composition assessment — Body composition assessment will be carried out using the BIA method on an eight-electrode body composition analyzer from TAnita. They will be marked:
  total mass, Total fat mass (FM) and segmental fat mass for five body segments: right leg (RL FM), Left leg (LL FM), right arm (RA FM), Left Arm (LA FM) trunk (TR FM).
  total fat-free mass (FFM) and segmental for five body segments: right leg (RL FFM), Left leg (LL FFM), right arm (RA FFM), Left Arm (LA FMM) trunk (TR FMM).
  Predicted total and segmental muscle mass (PMM) for five body segments: right leg (RL PMM), Left leg (LL PMM), right arm (RA PMM), Left Arm (LA PMM) trunk (TR PMM).
  Total water content (TBW) including intracellular water (ICW) and extracellular water (ECW)
  Groups: Adult group; Pediatric older group; School group; Senior group; Youth group
Diagnostic Test: assessment of body posture using the Kasperczyk method — The Kasperczyk method was used to assess body posture, including physiotherapeutic assessment in both standing and sitting positions. The symmetry of the head, shoulders, spine curvatures, knee joints and foot positioning were assessed. The symmetry of the head position was examined in all three planes and in all movements, i.e. flexion - extension, right turn - left turn, rotation and combined movements. The lateral curvatures of the spine (scoliosis) and their physiological curvatures, their deepening or shallowing in all sections of the spine, as well as the mobility of the spine in all physiological planes of movement were assessed. The position of the shoulder and hip girdle was assessed, as well as the position of the upper limbs at the level of the knees and feet. The mobility of the lower and upper limbs was examined.
  Groups: Pediatric group; Pediatric older group; School group; Senior group; Youth group
Diagnostic Test: Assessment of physical fitness — It depends on the age of the person being examined. In the case of children, the EUROFIT physical fitness test is carried out with modifications for age and gender. For the senior group, the Rikli and Jones test is used
  Groups: Adult group; Pediatric older group; School group; Senior group; Youth group
Diagnostic Test: Balance assessment — Balance assessment using the Zebris platform Static measurement - with eyes open and closed, assessing the load on the limbs during standing expressed in %, Balance analysis measurement - with eyes open and closed, test in a standing position, barefoot. The measurement duration is 30 seconds and the break between measurements is 30-60 seconds.
  Deflections of the center of gravity in the frontal and sagittal planes Length of the center of gravity swing path CoP - SPL [cm]. Inside the calculated ellipse lies 95% of the CoP location measurement data: amplitude, amplitude height, ellipse area (orientation of the direction of the ellipse's longitudinal axis relative to the platform's longitudinal axis, indicating clockwise rotation).
  Groups: Adult group; Pediatric older group; School group; Senior group; Youth group

SUMMARY:
The main aim of the research is to assess the impact of various forms of physical activity on body composition and posture. The basis of the research is the assessment of the current condition of people of different ages and the development of individualized physioprophylaxis programs for body posture and body weight abnormalities. In the senior group, the task of physioprophylactic programs is to prevent the loss of muscle mass, prevent falls and improve the quality of life.

DETAILED DESCRIPTION:
The research is focused on three age groups: research in the progressive period of ontogenesis from 3 to 18 years of age, people in adulthood, and people in senior age, i.e. postmenopausal women and men over 65 years of age. The research is conducted in three stages - in the first stage: assessment of the current condition, i.e. body weight and composition, assessment of body posture, physical fitness (including age-appropriate tests), assessment of physical activity (IPAQ test, PAQ-C and PAQ-A test). ). In the second stage: development and implementation of physioprophylactic programs aimed at preventing overweight or obesity, body posture abnormalities, and reduced physical fitness. Physioprophylactic projects based on medical training are adapted to age and gender and the assessment of the current condition. The duration of the training project is 12 weeks, classes will be held twice a week for 60 minutes for adults, twice a week for 45 minutes for children over 7 years of age and twice a week for 30 minutes for preschool children. Physioprophylactic classes will complement school classes for the group under 18 years of age. The third part of the research project is the assessment of changes in body weight, body posture and physical fitness.

The practical part will be complemented by meetings and lectures for the respondents and their parents (in the case of children) regarding the importance of physical activity, diet and physical fitness in the quality of life and its importance in various periods of ontogenetic development.

The study of a given group will be completed with a follow-up study 6 months after the end of the research project The ongoing research project will allow the development of physioprophylactic programs with elements of medical training to counteract lifestyle diseases.

ELIGIBILITY:
Inclusion Criteria:

* Informed written consent to participate in research and physical activity project of the examined person or his/her parent or legal guardian
* There are no health contraindications to physical activity
* no contraindications to the use of the bioelectrical impedance method (pacemaker, active cancer, pregnancy, metal elements in the body)

Exclusion Criteria:

* Remaining under the care of the Awad Postway correction clinic active therapeutic process of weight reduction
* being under the care of a cardiology clinic due to heart and/or circulatory system diseases - high blood pressure
* Condition after injuries to the spine,
* Orthopedic equipment - orthoses, prostheses, splints, crutches, walking aids
* lack of contact with the patient, impaired cognitive functions, inability to understand instructions when working in a group
* Diseases of the central nervous system
* Parkinson's disease, advanced senile dementia

Max Age: 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: The study group will be recruited from people living in the city of Wrocław and Lower Silesia from primary medical care centers, educational centers - kindergartens, and randomly selected primary schools. The Adult Group consists of people attending randomly selected secondary schools and various universities. The ej group will also include non-students recruited by invitation to participate in the research. The group of adults consists of people recruited on the basis of an open invitation carried out via social media, health facilities and large workplaces. The senior group will be recruited on the basis of an invitation addressed to senior activation centers
Sampling Method: Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2023-01-15 (Actual); Primary Completion 2028-12-31 (Estimated); Study Completion 2029-12-31 (Estimated)

PRIMARY OUTCOMES:
A physioprophylactic program for children aimed at normalizing body weight, improving physical fitness and correcting body posture | 01.2027-12.2027
  The result of the project will be the development of physioprophylactic programs based on medical training aimed at normalizing body weight, improving and correcting body posture and improving physical fitness. The programs will be adapted to the problems diagnosed in control tests and the age and gender of the examined children and adolescents Their final effectiveness will be assessed during follow-up tests performed immediately after the end of the 12-week program and follow-up tests after 6 months.
Physiophylaxis in adulthood | 01.2026-06.2027
  The result of the preliminary tests will be an estimate of the scale of occurrence of body weight abnormalities and body posture abnormalities, which are not monitored during this period. An important cognitive element will also be the assessment of the physical fitness of adults, taking into account their age, gender, body weight, forms of work undertaken, and exposure to stress.
  Their final effectiveness will be assessed during follow-up tests performed immediately after the end of the 12-week program and follow-up tests after 6 months.
Physiophylaxis in seniors | 01.2028-12.2028
  The result of the preliminary tests will be an estimate of the scale of occurrence of body weight abnormalities and body posture abnormalities, which are not monitored during this period. The physioprophylactic programs carried out will enable the development of standardized training programs aimed at improving the elderly's physical fitness, preventing falls, and maintaining the functionality and independence of older people. An important cognitive element will also be the assessment of the physical fitness of seniors, taking into account their age, gender, body weight, previously undertaken forms of work, exposure to stress, and quality of life.
  Their final effectiveness will be assessed during follow-up tests performed immediately after the end of the 12-week program and follow-up tests after 6 months.

CONTACTS AND LOCATIONS:
Overall Officials: AGNIESZKA CHWAŁCZYŃSKA, PROF, Principal Investigator — Wroclaw Uniwersity of Health and Sport Sciences
Locations (1):
- Faculty of Physiotherapy, Department of Human Biology, Wroclaw, Lower Silesian Voivodeship, Poland

IPD SHARING:
Plan to Share IPD: Undecided